CLINICAL TRIAL: NCT03640845
Title: Impact of a Hospital Medication Expertise on the Rate of Unplanned Hospitalizations at 3 Months of Patients Residing in Nursing Homes (EPAD)
Brief Title: Impact of a Hospital Medication Expertise on Unplanned Hospitalizations at 3 Months of Nursing Homes Patients
Acronym: TEM-EHPAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-16
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Age Problem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patient living in nursing homes a tele-expertise will be performed
  Interventions: Other: tele-expertise
- control group (No Intervention): Patient living in nursing homes will performed a normal care.

INTERVENTIONS:
Other: tele-expertise — Tele-expertise consists of the remote realization of a multi-professional medication review (clinical pharmacist and doctor / geriatrician), ie a complete and systematic analysis of sociodemographic, clinical, biological and pharmaceutical data transmitted in such a way standardized at the EHMP and aimed at optimizing the therapeutics of the resident patient of the EHPAD requesting tele-expertise.
  Tele-expertise is realized in three stages, that are
  * the transmission, the collection and the organization of the data,
  * the analysis of the data and their confrontation with the referential and recommendations
  * the writing of a Personalized Pharmaceutical Plan
  Arms: experimental group

SUMMARY:
The use of drugs in the elderly population remains a major public health problem worldwide. Technological advances and the development of new drugs have helped to extend life expectancy. However, the complex process of aging, resulting in changes in physiological functions, may affect the pharmacodynamics and kinetics of medications taken by the elderly. In addition, polypharmacy, due to multiple comorbidities, may also lead to an increased risk of drug or field interaction and the use of potentially inappropriate drugs (PID), increasing the risk of drug iatrogenic use in older users.

With a view to optimizing drug prescriptions and preventing drug iatrogenic disease in the elderly, and in the context of a university-based research and teaching approach, the AP-HM pharmacy initiated the setting up of clinical pharmacy activities for patients at high iatrogenic risk.

The contribution of clinical pharmacists to mobile geriatric teams who carry out more than 2,200 geriatric assessments a year, is a way to optimize the efficiency of the medication management of the elderly person hospitalized out of hospital. geriatric service and EHPAD. TIn order to promote the physician-pharmacist action synergy observed in practice, the investigators decided to integrate the pharmaceutical evaluation with the geriatric evaluation. This new cooperation makes it possible to improve the knowledge of the treatments taken by the patients, to raise awareness on the observance of the treatments and to facilitate the administration of the drugs, to reduce the risks of iatrogenic medicinal increase the acceptance of therapeutic interventions by the health care team. Indeed, the first results show that the mobile team's medico-pharmaceutical interventions have a much higher acceptance rate than medical or pharmaceutical interventions alone.

However, the economic context and the human resources allocated do not make it possible to ensure an efficient service throughout the territory and in particular in nursing homes outside the city where the CHU is located. In order to increase the number of evaluations, the investigators propose to develop a tele-expertise of a medico-pharmaceutical hospital team (MPHT) and evaluate the impact for patients residing in nursing homes in the context of a high-level study.

DETAILED DESCRIPTION:
The use of drugs in the elderly population remains a major public health problem worldwide. Technological advances and the development of new drugs have helped to extend life expectancy. However, the complex process of aging, resulting in changes in physiological functions, may affect the pharmacodynamics and kinetics of medications taken by the elderly. In addition, polypharmacy, due to multiple comorbidities, may also lead to an increased risk of drug or field interaction and the use of potentially inappropriate drugs (PID), increasing the risk of drug iatrogenic use in older users.

With a view to optimizing drug prescriptions and preventing drug iatrogenic disease in the elderly, and in the context of a university-based research and teaching approach, the AP-HM pharmacy initiated , in collaboration with certain clinical departments, the setting up of clinical pharmacy activities for patients at high iatrogenic risk. These activities were established and formalized in close collaboration with the doctors of the departments concerned, the geriatrics center and the geriatric mobile teams in particular, and were the subject of specific funding within the framework of the Instruction N ° DGOS / PF2 / 2016/49 of the 19/02/2016 relating to the call for project of implementation of the clinical pharmacy in health facility.

The contribution of clinical pharmacists to mobile geriatric teams (intra-hospital and outpatient), who carry out more than 2,200 geriatric assessments a year, is a way to optimize the efficiency of the medication management of the elderly person hospitalized out of hospital. geriatric service and EHPAD. In order to promote the physician-pharmacist action synergy observed in practice, the investigators decided to integrate the pharmaceutical evaluation (medication review) with the geriatric evaluation. This new cooperation makes it possible to improve the knowledge of the treatments taken by the patients, to raise awareness on the observance of the treatments and to facilitate the administration of the drugs (choice of the adapted galenic forms), to reduce the risks of iatrogenic medicinal increase the acceptance of therapeutic interventions by the health care team (attending physician, coordinator, nurse). Indeed, the first results show that the mobile team's medico-pharmaceutical interventions have a much higher acceptance rate than medical or pharmaceutical interventions alone.

However, the economic context and the human resources allocated do not make it possible to ensure an efficient service throughout the territory and in particular in nursing homes outside the city where the CHU (Marseille) is located. In order to increase the number of evaluations, the investigators propose to develop a tele-expertise of a medico-pharmaceutical hospital team (EHMP) and evaluate the impact for patients residing in nursing homes in the context of a high-level study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 65
* Resident in EHPAD
* presenting a high iatrogenic drug risk (Trivalle score between 6-10).
* Ability to provide free, informed and express consent (patient and / or trusted person)
* Affiliated to a social security scheme

Exclusion Criteria:

* Patient with a life expectancy <3 months
* Patient under 65 years
* Trivale score <6
* Vulnerable persons within the meaning of French law (adults under guardianship or trusteeship, persons deprived of their liberty)
* Participation in another research protocol in progress
* Patient who has had a medication review (or medication review) known in the last 6 months.
* Patient with severe dementia (MMSE <18)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2025-03-16 (Estimated); Study Completion 2025-09-16 (Estimated)

PRIMARY OUTCOMES:
number of unplanned hospitalizations | 6 months
  The main endpoint is the rate of unplanned hospitalizations (all structures) of nursing home residents

SECONDARY OUTCOMES:
Assessment of unplanned hospital admission | 6 months
  Number of unplanned hospital admissions
Quality of life (QoL) of nursing home residents | 3 months
  evaluated by the EuroQol 5-Dimension 3-Level (EQ-5D-3L) generic quality-of-life questionnaire. The EQ-5D-3L questionnaire will be administered (min 11111 - max 33333)
Quality of life (QoL) of nursing home residents | 6 months
  evaluated by the EuroQol 5-Dimension 3-Level (EQ-5D-3L) generic quality-of-life questionnaire. The EQ-5D-3L questionnaire will be administered (min 11111 - max 33333)
Incidence of behavioral disturbances | 3 months
  assessed by the NeuroPsychiatric Inventory (NPI) questionnaire. The total NPI score is the sum of the subscale scores (min 0 - max 120).
Incidence of behavioral disturbances | 6 months
  assessed by the NeuroPsychiatric Inventory (NPI) questionnaire. The total NPI score is the sum of the subscale scores (min 0 - max 120).
Proportion of residents subjected to at least 1 potentially inappropriate prescription | 3 months
  STOPP and START tool will be used for explicit criteria (French version 2).
Proportion of residents subjected to at least 1 potentially inappropriate prescription | 6 months
  STOPP and START tool will be used for explicit criteria (French version 2).
Nursing staff satisfaction with oral medications dispensed | 3 months
  Satisfaction is evaluated using 5-point Likert scales (Very satisfied - Satisfied - neutral - Dissatisfied - Very Dissatisfied)
Fall rate | 3 months
  Number of falls
Fall rate | 6 months
  Number of falls
Acceptation rate of general physician to therapeutic recommandations | 3 months
  Proportion of therapeutic recommendations accepted by general physician
Acceptation rate of general physician to therapeutic recommandations | 6 months
  Proportion of therapeutic recommendations accepted by general physician
Residents with at least 1 potentially inappropriate prescription | 3 months
  STOPP and START tool is used for explicit criteria (French version 2). The implicit approach includes all available medical data, potential self-medication, and questions from the Medication Appropriateness Index
Residents with at least 1 potentially inappropriate prescription | 6 months
  STOPP and START tool is used for explicit criteria (French version 2). The implicit approach includes all available medical data, potential self-medication, and questions from the Medication Appropriateness Index
Description of patients whose general physician have taken account of recommendations | 3 months
  Demographics, diseases, medications and types of recommendations made from patients for whom at least 50% of recommendations have been accepted
Characteristics of patients whose GP have taken account of TMR recommendations | 3 months
  : Demographics, diseases, medications and types of recommendations made from patients for whom at least 50% of recommendations have been accepted
Incremental cost-effectiveness ratio | 6 months
  Incremental cost-effectiveness ratio (ICER) is used to compare the cost effectiveness of the experimental strategy with that of standard care. It is the ratio of the difference in costs between groups to the difference in effectiveness
Qualitative acceptability intervention survey | 6 months
  Intervention acceptability survey is carried out to determine care provider acceptance and expectations of intervention in nursing homes.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, MD, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France

REFERENCES:
- [Derived] Berard C, Di Mascio T, Montaleytang M, Couderc AL, Villani P, Honore S, Daumas A, Correard F. Telemedication Reviews to Optimize Medication Prescription for Older People in Nursing Homes. Telemed J E Health. 2022 Aug;28(8):1225-1232. doi: 10.1089/tmj.2021.0288. Epub 2021 Dec 24. PMID 34958258
- [Derived] Correard F, Montaleytang M, Costa M, Astolfi M, Baumstarck K, Loubiere S, Amichi K, Auquier P, Verger P, Villani P, Honore S, Daumas A. Impact of medication review via tele-expertise on unplanned hospitalizations at 3 months of nursing homes patients (TEM-EHPAD): study protocol for a randomized controlled trial. BMC Geriatr. 2020 Apr 20;20(1):147. doi: 10.1186/s12877-020-01546-3. PMID 32312242